CLINICAL TRIAL: NCT02843243
Title: A Prospective, Multicenter Validation of Different Risk Assessment Strategies in Normotensive Patients With Acute Pulmonary Embolism
Brief Title: Validation of Different Risk Assessment Strategies in Normotensive Pulmonary Embolism
Status: Terminated | Type: Observational
Why Stopped: slow recruitment rate. new study planned
Sponsor: Azienda Ospedaliera Cosenza (Other)
Responsible Party: Sponsor
Other Study IDs: bova 1 protocol
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A risk stratification in hemodynamically stable patients with acute pulmonary embolism (PE) is deemed necessary to guide patient management. With the aim to improve the positive predictive value (PPV) for PE-related adverse events in in normotensive patients, a number of scores combining multiple risk-factors have been published. In addition, an algorithm for the risk-stratification of patients with PE has been proposed by the European society of cardiology. None but one of these scores underwent external and prospective validation. The aim of this study is to externally and prospectively validate the PPV for PE-related adverse events of the Bova score and modified FAST score in a large multicenter cohort.

DETAILED DESCRIPTION:
A risk stratification in hemodynamically stable patients with acute pulmonary embolism (PE) is deemed necessary to guide patient management. Right ventricular dysfunction (RVD), identified by echocardiography or computed tomographic angiography (CT), and cardiac biomarkers are well recognized risk factors for adverse events in normotensive patients with PE. However, neither of them, as a single prognostic criterion, have a sufficient positive predictive value (PPV) for PE-related adverse events to guide therapeutic decisions. The PEITHO trial showed that, in normotensive patients with RVD and abnormal cardiac troponin, death or hemodynamic decompensation occurred significantly less in those treated with tenecteplase plus heparin than in those who received heparin plus placebo. However the risk of major hemorrhage and stroke was significantly increased in the tecneplase group. These results were obtained in a group of patients with an absolute rate of PE-related adverse events of about 6%. If the same relative reduction in the risk of PE-related outcomes observed in the PEITHO trial could be achieved in a group of patients with a higher absolute risk of PE-related events, this might change the risk to benefit ratio of primary reperfusion therapy in PE. With the aim to improve the PPV for PE-related adverse events in in normotensive patients, a number of scores combining multiple risk-factors have been published. In addition, an algorithm for the risk-stratification of patients with PE has been proposed by the European society of cardiology. None but one of these scores underwent external and prospective validation. Aim of the study The aim of this study is to externally and prospectively validate the PPV for PE-related adverse events of the Bova score, modified FAST score and ESC algorithm in a large multicenter cohort.

Methods. This will be a multicenter, prospective, observational study. Consecutive patients aged 18 years or older with PE and hemodynamic stability (that is, SBP 90 mm Hg or more) will be evaluated as a part of usual clinical practice. This study does not dictate diagnostic interventions nor affects clinical or therapeutic decisions of the participant centers. For each patient, anonymous information will be collected on simplified Pulmonary Embolism Severity Index (sPESI), RVD on echocardiography and CT, Troponin I, levels of lactates in the arterial blood, and presence of syncope at presentation. RVD will be diagnosed with the echocardiography in the presence of one of the following: Right ventricular end-diastolic diameter (RVEDD) > 30 mm (parasternal long-axis or short-axis view), Right/left ventricular end-diastolic diameter (RVEDD/LVEDD) >0.9 (apical or subcostal 4-chamber view), Right ventricular free wall hypokinesis from any view, Tricuspid systolic velocity > 2.6 m/s from the apical or subcostal 4-CH view, parasternal short-axis view. RVD diagnosis with the CT will require a RV/LV diameter ratio greater than 1.0 on axial CT images. Cardiac troponin test will be considered positive in case of levels of troponin higher than higher than the cut-off of the manufacturer. Plasma lactate will be assessed in arterial blood samples. Values ≥ 2 mmol/L (18 mg/dL) will be considered abnormal. This evaluation should be ideally completed within 6 hours from the hospital admission. The primary outcome of the study will be adverse events PE-related within 30 days from the hospital admission. In a sensitivity analysis we will explore the same outcome at 7 days. PE-relate adverse events will be defined as: PE-related death or haemodynamic collapse. PE will be considered the cause of death if there will be objective documentation or in case of unexplained death and PE not confidently ruled out. Haemodynamic collapse will be defined as one of the following conditions: SBP < 90 mmHg necessitating catecholamine administration; mechanical ventilation; cardiopulmonary resuscitation.

Secondary outcomes of interest will be all-cause mortality at 30 days; PE-related death at 30 days; confirmed symptomatic PE recurrence; duration of hospitalization in patients with low and intermediate-low risk compared with patients with intermediate-high risk. Recurrent PE will be confirmed either by the presence of a new intraluminal filling defect, or by a new perfusion scan defect involving > 75% of a lung segment. PE-related adverse events, recurrent PE and all-cause mortality should be evaluated, for each participant center, by a physician not involved in the study.

Statistical analysis The three-level of Bova score will be dichotomized (low- and intermediate-low-risk versus intermediate-high-risk). Receiver operating characteristic (ROC) curve analysis will be performed to determine the area under the curve (AUC) of the scores (absolute points) with regard to study outcomes. Prognostic performance of the scores will be evaluated by calculation of sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV), and positive and negative likelihood ratios.

Sample size Based on previous studies a sample size of about 500 patients should be adequate for the purpose of the study. After the first 300 patients an interim analysis will be performed to more precisely establish the number of patients needed.

ELIGIBILITY:
Inclusion Criteria:

Pulmonary Embolism with hemodynamic stability (that is, SBP 90 mm Hg or more)

Exclusion Criteria:

Refuse of informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients aged 18 years or older with Pulmonary Embolism and hemodynamic stability (that is, SBP 90 mm Hg or more)
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-12; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse events PE-related | within 30 days from the hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Bova, MD, Principal Investigator — Azienda Ospedaliera Cosenza
Locations (1):
- Azienda ospedaliera Cosenza, Cosenza, Italy

IPD SHARING:
Plan to Share IPD: Yes